CLINICAL TRIAL: NCT06511635
Title: Multicenter Quantitative and Qualitative Study of the Determinants of Participation in a Cytomegalovirus Preventive Vaccine Study in France in Women Aged 18 to 40 Years Old.
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN432024/CHUSTE
Record Dates: First submitted 2024-07-09; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Recruitment
Keywords: Recruitment methods; Determinants; CMVCTORY vaccine trial; women's participation; vaccine trial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women between 18 to 40 included in CMVCTORY vaccine trial: Women between 18 to 40 included in CMVCTORY vaccine trial will be included.
  Interventions: Other: Qualitative interview; Other: Quantitative questionnaire

INTERVENTIONS:
Other: Qualitative interview — Interview between participant and a researcher, in order to identity the determinants of participation in a clinical trial among participants in the CMVictory vaccine trial.
Other: Quantitative questionnaire — Anonymous online survey using a 3-part questionnaire, studying knowledge of clinical research and the determinants of participation in a preventive vaccine study in a population of young women (aged 18-40).

SUMMARY:
During a vaccine clinical trial of Cytomegalovirus (CMV) vaccine, one of the participants' motivations was to prevent an infection responsible for malformations in a future child. Would their attitude towards a vaccine trial be the same in the context of a vaccine designed to protect them individually? By improving the knowledge of clinical research and determinants in women aged 18 to 40, this study could improve recruitment methods in this specific population for future vaccine trials within the CIC1408 infectious diseases and vaccinology area at Saint-Etienne University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Womens between 18 to 40 included in CMVCTORY vaccine trial

Exclusion Criteria:

* Refusal

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All french participants of the CMVCTORY vaccine trial.
Sampling Method: Non-Probability Sample
Enrollment: 306 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
qualitative interview | Day : 1
  To identify the motivations and the obstacles of participation in an experimental trial in women of childbearing age in Phase 3 trial.

CONTACTS AND LOCATIONS:
Overall Officials: Nelly JACQUEMET, nurse, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Centre Hospitalier Universitaire de St Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No